CLINICAL TRIAL: NCT03990168
Title: The Effect of the Combined Treatment Approach of Delayed Auditory Feedback and Transcranial Direct Current Stimulation to Enhancement of Speech Fluency in Adults Who Stutter
Brief Title: The Effect of the Non-invasive Brain Stimulation on the Speech Fluency Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Moin, Principal Investigator, Iran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 98-2-75-15001
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Stuttering/ Developmental
MeSH Terms: conditions — Stuttering | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will receive one anodal tDCS at 1 mA intensity over the left superior temporal gyrus (T3 in 10-20 international system) and the cathode tDCS over the right orbitofrontal area (Fp2 in 10-20 international system). tDCS will be delivered for 20 minutes during fluency intervention for six consecutive days.
  Interventions: Device: Anodal tDCS; Behavioral: fluency intervention/ Delayed Auditory Feedback
- Sham Comparator (Sham Comparator): Participants will receive sham tDCS while the one anode electrode will be positioned over the left superior temporal gyrus and the cathode will be placed over the right orbitofrontal similar to the active mode. The sham stimulation will break down after 30 seconds at the beginning of 20 minutes of fluency intervention for six consecutive days.
  Interventions: Behavioral: fluency intervention/ Delayed Auditory Feedback; Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — 1 mA anodal tDCS positioned over left superior temporal gyrus and the cathode placed over the occipital lobe. The tDCS stimulation will be delivered for 20 minutes on 6 intervention days.
  Arms: Experimental
Behavioral: fluency intervention/ Delayed Auditory Feedback — Each participant complete three tasks include reading, conversation, and narration. Delayed auditory feedback will be used during these tasks. Each treatment session will take 20 minutes.
Device: Sham tDCS — The anodal tDCS positioned over left superior temporal gyrus and the cathode placed over the occipital lobe. The current of sham stimulation will involve 30 seconds of stimulation at the beginning of the 20 minutes on 6 intervention days.
  Arms: Sham Comparator

SUMMARY:
The aim of this study is to determine the effectiveness of concurrent transcranial direct current stimulation (tDCS) and fluency training in adults with developmental stuttering. We examine the severity of stuttering to investigate the effect of treatnment. In the control group the anodal tDCS and DAF will applied on six consecutive days (1 milliampere [mA] for 20 mins per day), and the control group will received the sham stimulation and DAF for the same time. The severity of stuttering measured by means of tasks and questionnaires before and after treatment sessions and 6 weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of developmental stuttering
* Participants diagnosed with moderate to severe stuttering
* Right handed
* Native speaker of Farsi

Exclusion Criteria:

* Speech or language disorders other than stuttering
* Received stuttering treatment within the past year
* Hearing loss
* History of neurological or psychiatric disorders
* History of seizure
* Taking any medication that may affect brain function such as anti-depressants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Mean score of percentage of Stuttered Syllables produced in the speech sample | Baselines, immediately post-treatment, 1-week post-treatment, 6-weeks post-treatment
  Researcher will calculate the Percentage of Stuttered Syllables (SS %) in the speech sample. Lower percentage of Stuttered Syllables represents better outcomes.

SECONDARY OUTCOMES:
Mean score of the Stuttering Severity Instrument version 4 (SSI-4) | Baselines, immediately post-treatment, 1-week post-treatment, 6-weeks post-treatment
  The Stuttering Severity Instrument (SSI-4) is a standardized measure of stuttering severity consist of of 3 subscales (frequency, duration and physical concomitants) which are summed to give a total score. The maximum total score of the SSI-4 is 56, which corresponds to the highest stuttering severity. So, lower score represents better outcomes.
Mean score of the Overall Assessment of Speakers Experience of Stuttering (OASES) | Baselines, immediately post-treatment, 1-week post-treatment, 6-weeks post-treatment
  The OASES is a standardized assessment to measure the effect of stuttering on a person's life that consists of 4 subscales (general information about speech, your reactions to stuttering, communication in daily situations, quality of life). Each sub-test has a score from 1 to 5 in which the number 1 indicates the least negative impact and number 5 shows the most negative impact. These are combined to give a total impact score between 1 and 5, with 5 representing the highest negative impact on person's life. So, higher score represents better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Reyhane Mohamadi, Study Director — Iran University of Medical Sciences
Locations (1):
- Narges Moin, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moein N, Mohamadi R, Rostami R, Nitsche M, Zomorrodi R, Ostadi A, Keshtkar A. Delayed Auditory Feedback and Transcranial Direct Current Stimulation Treatment for the Enhancement of Speech Fluency in Adults Who Stutter: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Apr 21;9(4):e16646. doi: 10.2196/16646. PMID 32314973